CLINICAL TRIAL: NCT02753738
Title: Enhancement of Learning Associated Neural Plasticity by Selective Serotonin Reuptake Inhibitors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Prof MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21042016
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Ssri; Neuronal Plasticity
MeSH Terms: interventions — Escitalopram; Diffusion Tensor Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SSRI treatment (Experimental): Subjects will receive 21 days of 10mg escitalopram treatment while performing learning paradigms.
  Interventions: Drug: Escitalopram; Other: 3xMR scan (fMRI, DTI, strucutral MRI); Behavioral: Association learning paradigm; Behavioral: Association re-learning paradigm
- Placebo treatment (Placebo Comparator): Subjects will receive 21 days of placebo treatment while performing learning paradigms.
  Interventions: Drug: Placebo; Other: 3xMR scan (fMRI, DTI, strucutral MRI); Behavioral: Association learning paradigm; Behavioral: Association re-learning paradigm

INTERVENTIONS:
Drug: Escitalopram — Tablet 10mg, 21 days
  Arms: SSRI treatment
Drug: Placebo — Tablet, 21 days
  Arms: Placebo treatment
Other: 3xMR scan (fMRI, DTI, strucutral MRI) — 3 Tesla PRISMA MAGNETOM MR scanner; performed at baseline, after 21 days of performing learning paradigms and after 21 days of drug/placebo treatment and re-learning paradigms
Behavioral: Association learning paradigm — 21 daily internet-based sessions (20min) of learning associations (pairs) of stimuli
Behavioral: Association re-learning paradigm — 21 daily internet-based sessions (20min) of learning new associations (pairs) of stimuli performed during escitalopram/placebo treatment

SUMMARY:
Background:

Conclusive evidence states that the serotonergic system mediates neuroplasticity from early embryonic development until brain maturation in adulthood. This study aims to demonstrate that selective serotonin reuptake inhibitors (SSRIs) enhance learning-dependent neuroplasticity in vivo, hereby contributing to the investigators understanding of the mechanism of action of therapy with SSRIs.

Objectives:

1. To prove a positive influence of SSRIs on structural remodeling during learning, reflected by enhancements of gray and white matter microstructure, connectivity and functionality in brain regions involved in learning processes.
2. To show that this effect is topologically specific, i.e. that enhancements of plasticity markers are found in different regions depending on their involvement during the performance of specific learning tasks.

Study design:

Randomized, double-blind, placebo-controlled, longitudinal mono-center study. 80 healthy subjects will undergo three MRI scanning sessions: 1. baseline, at study entry, 2. after 3 weeks of facial/emotional (n=40) or Chinese character-meaning learning (n=40) and 3. after 3 weeks learning of new associations under administration of an SSRI or placebo.

Methods:

MRI measurements will be performed on a 3 Tesla PRISMA MAGNETOM MR scanner. Changes in gray matter microstructure will be assessed using high-resolution structural MRI and analyzed with voxel-based morphometry (VBM). Diffusion tensor imaging (DTI) enables non-invasive investigation of neuroplasticity in the human brain based on the reduction in mean diffusivity associated with swelling of astrocytes after increased synaptic activity. Resting-state functional MRI (fMRI) will allow for the measurement of changes in functional coupling between brain regions, and fMRI during tasks will assess differential activity in brain regions during learning.

Relevance and implications:

This study aims to provide evidence that SSRIs facilitate cytoarchitectonical restructuring. In addition to expanding the investigators current knowledge on the trophic effects of SSRIs, the results of this study will also elucidate interactions between the serotonergic system and changes to neuronal networks during learning as well as their behavioral consequences. By probing the neurobiological correlates of the antidepressant and anti-anxiety effects of SSRIs, this study will provide a rationale for targeted interventions that harness the neuroplasticity enhancing properties of SSRIs to facilitate therapeutic processes.

ELIGIBILITY:
Inclusion Criteria:

* General health based on medical history, physical examination and structured clinical interview for DSM-IV (SCID)
* Willingness and competence to sign the informed consent form
* Right-handedness
* Non-smoker, and non-alcohol drinker

Exclusion Criteria:

* Any medical, psychiatric or neurological illness
* Current or former substance abuse
* Any implant or stainless steel graft or any other contraindications for MRI
* First degree relatives with a history of psychiatric illness or substance abuse
* Color blindness, any Chinese language skills
* Failure to comply with the study protocol or to follow the instructions of the investigating team
* Lifetime use of SSRIs or related psychotropic agents
* Non-Caucasian

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Gray matter volume | 21 days
  voxel based morphometry (T1 weighted MPRAGE sequence)
Mean diffusivity | 21 days
  diffusion tensor imaging

SECONDARY OUTCOMES:
BOLD signal | 21 days
  functional MRI (learning paradigms)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Vanicek T, Reed MB, Seiger R, Godbersen GM, Klobl M, Unterholzner J, Spurny-Dworak B, Gryglewski G, Handschuh P, Schmidt C, Kraus C, Stimpfl T, Rupprecht R, Kasper S, Lanzenberger R. Increased left dorsolateral prefrontal cortex density following escitalopram intake during relearning: a randomized, placebo-controlled trial in healthy humans. Ther Adv Psychopharmacol. 2022 Nov 17;12:20451253221132085. doi: 10.1177/20451253221132085. eCollection 2022. PMID 36420117
- [Derived] Vanicek T, Reed MB, Unterholzner J, Klobl M, Godbersen GM, Handschuh PA, Spurny-Dworak B, Ritter V, Gryglewski G, Kraus C, Winkler D, Lanzenberger R, Seiger R. Escitalopram administration, relearning, and neuroplastic effects: A diffusion tensor imaging study in healthy individuals. J Affect Disord. 2022 Mar 15;301:426-432. doi: 10.1016/j.jad.2021.12.135. Epub 2022 Jan 10. PMID 35016914